CLINICAL TRIAL: NCT02988700
Title: Safety and Analgesic Efficacy of Spinal Versus Caudal Block in Pediatric Infra-umbilical Surgery
Brief Title: Spinal Versus Caudal Analgesia After Pediatric Infra-umbilical Surgery
Acronym: ITVSEpidural
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Assisstant professor in anesthesia and intensive care, Faculty of medicine, Assiut university, Egypt., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008718/36800
Record Dates: First submitted 2016-11-25; First posted 2016-12-09 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; bucain

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal group (Active Comparator): Intrathecal hyperbaric bupivacaine 0.25mg/kg will be give by lumber puncture that will be made in the lateral position at the L4-5 or L5-S1 interspace with a 25 G pencil point Quincke spinal needle with a short bevel and the orifice of the spinal needle will be turned cephalad.
  be given by .
  Interventions: Drug: Intrathecal hyperbaric bupivacaine 0.25mg/kg 0.5%
- Caudal group (Active Comparator): caudal plain bupivacaine 2.5mg/kg 0.25% will be given caudally in The sacral hiatus between the sacral conru that will be palpated. While inserting the 23-G needle at 45° to the skin in the midline, a distance "give" or "pop" will be felt as the needle passes the sacral ligament into the caudal space, the needle will be tilted more toward the skin surface and inserted 2-3mm deeper.
  Interventions: Drug: caudal plain bupivacaine 2.5mg/kg 0.25%

INTERVENTIONS:
Drug: Intrathecal hyperbaric bupivacaine 0.25mg/kg 0.5% — The lumber puncture will be made in the lateral position at the L4-5 or L5-S1 interspace with a 25 G pencil point Quincke spinal needle with a short bevel and the orifice of the spinal needle will be turned cephalad.
  Other Names: Marcain
  Arms: Spinal group
Drug: caudal plain bupivacaine 2.5mg/kg 0.25% — The sacral hiatus between the sacral conru will be palpated. While inserting the 23-G needle at 45° to the skin in the midline, a distance "give" or "pop" will be felt as the needle passes the sacral ligament into the caudal space, the needle will be tilted more toward the skin surface and inserted 2-3mm deeper.
  Other Names: Bucain
  Arms: Caudal group

SUMMARY:
Caudal analgesia along with general anesthesia is a very popular regional technique for prolonged postoperative analgesia in different pediatric surgical procedures where the surgical site is sub-umbilical. Caudal anesthetics usually provide analgesia for approximately 4-6 hours.

Recently, the use of spinal anesthesia in infants and children requiring surgeries of sub-umbilical region is gaining considerable popularity worldwide.

- The ease of performance and the safety regarding cardio-respiratory functions makes spinal anesthesia as an alternative to general anesthesia in infants and children undergoing surgeries of sub-umbilical regions.

DETAILED DESCRIPTION:
The historic view that young children neither respond to, nor remember, painful experiences to the same degree as adults is no longer thought to be true. About 40% of pediatric surgical patients experienced moderate or severe postoperative pain and 75% had insufficient analgesia.

-Pediatric acute pain services use techniques of concurrent or co-analgesia based on four classes of analgesics, namely local anesthetics, opioids, non-steroidal anti-inflammatory drugs (NSAIDs), and acetaminophen (paracetamol).

Caudal analgesia along with general anesthesia is a very popular regional technique for prolonged postoperative analgesia in different pediatric surgical procedures where the surgical site is sub-umbilical. Caudal anesthetics usually provide analgesia for approximately 4-6 hours.

Recently, the use of spinal anesthesia in infants and children requiring surgeries of sub-umbilical region is gaining considerable popularity worldwide.

- The ease of performance and the safety regarding cardio-respiratory functions makes spinal anesthesia as an alternative to general anesthesia in infants and children undergoing surgeries of sub-umbilical regions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-12 years.
* Weight: 15-40 kg.
* Sex: both males and females.
* ASA physical status: 1-II.
* Operation: surgery below umbilicus.

Exclusion Criteria:

* Allergic reaction to local anesthetics (LAs).
* Local or systemic infection (risk of meningitis).
* Coagulopathy.
* Intracranial hypertension.
* Hydrocephalus.
* Intracranial hemorrhage.
* Parental refusal.
* Hypovolemia.
* Spinal deformities, such as spina bifida or myelomeningocele.
* Presence of a ventriculoperitoneal shunt because of a risk of shunt infection or dural leak.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-11; Primary Completion 2018-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
FLACC Score | 24 hours
  FLACC scores will be recorded.

SECONDARY OUTCOMES:
Total consumption of rescue analgesics | 24 hours
  The total consumption of postoperative rescue analgesics will be recorded.
Postoperative Agitation | 60 min.
  Postoperative agitation will be evaluated by the Four Point Agitation Sedation scale.
Adverse effects | 24 hours
  Any adverse effect will be treated and recorded.
Residual motor paralysis | 6 hours
  By the Modified Bromage scale

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assisstant professor in anesthesia and intensive care, faculty of medicine, Assiut university, Egypt
Locations (1):
- Hala Saad Abdel-Ghaffar, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No